CLINICAL TRIAL: NCT02066272
Title: Safety of Anti-TNF Antibodies, Including Biosimilars, in Treatment of Inflammatory Bowel Disease: Multicentre Cohort Observational Study (SATIMOS)
Brief Title: Safety of Anti-tumor Necrosis Factor (TNF) Monoclonal Antibodies in Inflammatory Bowel Disease
Acronym: SATIMOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: The Children's Memorial Health Institute, Poland (Unknown); Intestinal Section of the Polish Society of Gastroenterology (Unknown)
Responsible Party: Principal Investigator, Edyta Zagorowicz, MD, PhD, Maria Sklodowska-Curie National Research Institute of Oncology
Other Study IDs: 29/2013
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease; Indeterminate Colitis
Keywords: IBD; anti-TNF; biosimilars; safety
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IBD patients: IBD patients who start or re-start anti-TNF therapy

SUMMARY:
Anti-TNF (tumor necrosis factor) monoclonal antibodies have revolutionized management of Inflammatory bowel disease. Their common features include high efficacy but also immunogenicity and increased infection risk. Since 2013, two generics or biosimilars of the first anti-TNF have been registered in Europe, which long lerm safety profile needs yet to be established.

This prospective, multicenter, observational cohort study will assess safety of treatment of anti-TNF monoclonal antibodies in inflammatory bowel disease patients in Poland.

Eligible are consecutive patients in whom anti-TNF is started for Crohn's disease, ulcerative colitis or indeterminate colitis between January 1st, 2014 and December 31st, 2015. Data to be collected include demography, Montreal classification, indication to treatment, previous treatment, operations, extraintestinal manifestations and concomitant diseases. Data on response, tolerability and safety of anti-TNF and on concomitant treatment will be collected. Adverse events logs will be completed. Majority of IBD centres in Poland, pediatric and adult, academic and regional, have agreed to participate in the study.

As a result of the study, the frequency of adverse events in a cohort of Polish IBD patients on various anti-TNFs will be established.

DETAILED DESCRIPTION:
1. This is a prospective observational study aimed to register adverse events occuring on biological treatment in inflammatory bowel disease (IBD) patients in Poland.
2. Eligible are pediatric and adult patients in whom anti-TNF (tumor necrosis factor) treatment is started for Crohn's disease, ulcerative colitis or indeterminate colitis, financed by the National Health Care System and who gave their informed consent for participation in the study (for children the consent of a parent is required).
3. The study data are collected in a dedicated on-line data - base.
4. Each centre participating in the study is obliged to screen for the study all consecutive patients in whom the biological treatment is started. If a patient refuses to consent, this information must have been documented in the data - base.
5. Patient data collected at the start of anti-TNF treatment include the type of anti-TNF, demographic data, the type, extension or location, course and activity of IBD, indication to biological treatment, history of previous treatment, operations, extraintestinal manifestations and co-existing diseases. As regards to the anti-TNFs, biosimilars are categorised as distinct drugs in order to separately follow-up the safety profile of each.
6. Data on response, tolerability and safety of anti-TNF and on concomitant treatment are updated following each visit. Adverse events logs and serious adverse events log are completed if necessary.
7. Registration of new patients will be ongoing from Jan 2014 do Dec 2015. After this time, a centre may choose to continue doing the study.
8. In addition, data on health events in enrolled patients will be collected independently from the National Health Care System database, also after the on-site observation of patients is completed.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with pre-diagnosed ulcerative colitis, Crohn's disease or undeterminate colitis who start or re-start anti-TNF treatment in a study centre
* Gave their consent to participate in the study (in children, caretakers consent is required)

Exclusion Criteria:

* Lack of the patient's consent
* Participation in a clinical trial with anti - TNFs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All IBD patients who start or re-start anti-TNF therapy within the study period.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The frequency of adverse events on induction of remission and maintenance treatment using anti-TNFs (including biosimilars) in a cohort of IBD patients | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Edyta Zagorowicz, MD, PhD, Principal Investigator — Department of Gastroenterological Oncology, The Maria Sklodowska-Curie Memorial Cancer Centre and Institute of Oncology, Warsaw, Poland; Jaroslaw Kierkus, MD, PhD, Principal Investigator — Department of Gastroenterology, Hepatology and Feeding Disorders, The Children's Memorial Health Institute, Warsaw , Poland; Maria Klopocka, MD, PhD, Study Chair — Interventional Endoscopy Center, Outpatient Department for Bowel Diseases, University Hospital nr 2 in Bydgoszcz, Poland; Maria Wisniewska-Jarosinska, MD, PhD, Study Chair — Gastroenterology and Endoscopy Unit, Medical University of Lodz, St Family Hospital, Lodz, Poland
Locations (2):
- Poland (2):
  - Department of Gastroenterology and Hepatology, Medical Center for Postgraduate Education and The Maria Sklodowska-Curie Memorial Cancer Centre and Institute of Oncology, Warsaw, Masovian Voivodeship
  - Department of Gastroenterology, Hepatology and Feeding Disorders, The Children's Memorial Health Institute, Warsaw, Masovian Voivodeship